CLINICAL TRIAL: NCT02022215
Title: A Phase 2 Randomized, Double-Blind, Vehicle-Controlled, Dose-Ranging Study to Investigate the Efficacy and Safety of ME1111 in Patients With Mild to Moderate Onychomycosis
Brief Title: Efficacy and Safety Study of ME1111 in Patients With Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ME1111-2
Record Dates: First submitted 2013-12-15; First posted 2013-12-27 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ME1111 Solution, Low strength (Experimental)
  Interventions: Drug: ME1111 Solution, Low strength
- ME1111 Solution, High strength (Experimental)
  Interventions: Drug: ME1111 Solution, High strength
- Matching Vehicle Solution (Placebo Comparator)
  Interventions: Drug: Matching Vehicle Solution

INTERVENTIONS:
Drug: ME1111 Solution, Low strength — ME1111 Solution, Low strength, applied once daily for 48 weeks
  Arms: ME1111 Solution, Low strength
Drug: ME1111 Solution, High strength — ME1111 Solution, High strength, applied once daily for 48 weeks
  Arms: ME1111 Solution, High strength
Drug: Matching Vehicle Solution — Matching Vehicle Solution, applied once daily for 48 weeks
  Arms: Matching Vehicle Solution

SUMMARY:
The purpose of the study is to determine the safety and efficacy of high and low strength of ME1111 solutions compared to the vehicle in the treatment of onychomycosis of the toenail.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate distal lateral subungual onychomycosis
* A positive potassium hydroxide (KOH) microscopy
* A positive fungal culture for a dermatophyte
* Good general health

Exclusion Criteria:

* Uncontrolled diabetes
* Onychomycosis of the fingernails
* Prior use of antifungal drugs (Failure to complete the specified washout period)
* History of HIV, Hepatitis B or Hepatitis C
* Diagnosis of psoriasis or history of psoriasis
* Participated in any other trial of an investigational drug or device within 30 days or participation in a research study concurrent with this study
* Pregnancy/lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2015-10-28 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Complete cure rate at Week 52 | Week 52
  complete cure :clear (zero %) clinical involvement of the target great toenail and mycologic cure.

SECONDARY OUTCOMES:
Complete or almost complete cure rate at Week 52 | Week 52
  complete or almost complete cure:5 % or less clinical involvement of the target great toenail and mycologic cure.
Number of Adverse events | Up to Week 48, Week 52, EOS
Local Tolerability Assessments | Up to Week 48, Week 52, EOS
  Local Tolerability Assessments:Burning/Stinging, Pruritus, Dryness, Scaling, Erythema, General Irritation, Induration/Edema, Oozing/crusting.

CONTACTS AND LOCATIONS:
Overall Officials: Meiji Study Director, Study Director — Meiji Seika Pharma Co., Ltd.
Locations (31):
- United States (31):
  - Birmingham, Alabama
  - Encinitas, California
  - San Diego, California
  - San Francisco, California
  - Santa Rosa, California
  - Denver, Colorado
  - Miami, Florida
  - Miramar, Florida
  - Newnan, Georgia
  - Boise, Idaho
  - Evansville, Indiana
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Clinton Township, Michigan
  - Fridley, Minnesota
  - Albuquerque, New Mexico
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Mt. Pleasant, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Lynchburg, Virginia
  - Norfolk, Virginia
  - Spokane, Washington